CLINICAL TRIAL: NCT06194799
Title: A 52-Week, Open-Label Extension Study of ACP-204 in Adults With Alzheimer's Disease Psychosis
Brief Title: ACP-204 in Adults With Alzheimer's Disease Psychosis Open Label Extension Study
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-204-008; Luminous (Other: Acadia Pharmacueticals)
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer's Disease Psychosis
Keywords: Alzheimer's Disease Psychosis; Hallucinations; Delusions
MeSH Terms: conditions — Hallucinations; Delusions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACP-204 (Experimental): ACP-204 30mg or 60mg
  Interventions: Drug: ACP-204

INTERVENTIONS:
Drug: ACP-204 — ACP-204 30 mg given once daily, as capsule OR ACP-204 60 mg given once daily, as capsule

SUMMARY:
This 52-week, open-label extension study is to evaluate the long-term safety and tolerability of ACP-204 in subjects with ADP.

ELIGIBILITY:
Inclusion Criteria:

* Subject has successfully completed ACP-204-006 study
* Male or female (age 55 to 95 years old): female must be of non-childbearing potential, male must take appropriate contraceptive method if partner has childbearing potential
* Subject has a designated study partner/caregiver
* Subjects are able to complete all study visits with a study partner/caregiver
* Signed inform consent form with a caregiver or legal representative

Exclusion Criteria:

* Requires treatment with a medication prohibited by the protocol
* Is in hospice and receiving end-of-life palliative care, or has become bedridden
* Unstable clinically significant medical condition other than AD
* Any medical condition that in the opinion of the investigator may affect safety or ability to complete the study

Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | 52 Weeks
  Number of Subjects With Adverse Events (AEs), Discontinuations Due to AEs and Serious AEs (SAEs) over 52 weeks of treatment. The Safety population consists of all subjects who received at least one dose of study drug in this study.

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement in the ADP context (CGI-I-ADP) score | 52 Weeks

CONTACTS AND LOCATIONS:
Locations (65):
- United States (15):
  - ATP Clinical Research, Costa Mesa, California
  - New Life Medical Research Center, Hialeah, Florida
  - Reliable Clinical Research LLC, Hialeah, Florida
  - Homestead Associates in Research Inc., Miami, Florida
  - Premier Clinical Research Institute Inc, Miami, Florida
  - Advanced Clinical Research, Miami, Florida
  - Verus Clinical Research, Miami, Florida
  - Future Care Solution, LLC, Miami, Florida
  - MediClear Medical & Research Center, Inc., Miami, Florida
  - ABBA Medical Research LLC, Miami, Florida
  - New Med Research, Miami Gardens, Florida
  - Floridian Neuroscience Institute, Miami Lakes, Florida
  - Abington Neurological Associates, Abington, Pennsylvania
  - Uni Texas Health Science Center, Houston, Texas
  - Clinical Trial Network LLC, Houston, Texas
- Brazil (8):
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Universitario de Brasilia, Brasília
  - TrialTech Tecnologia com Pesquisas em Medicamentos, Curitiba
  - Inst de Neurologia de Curitiba Hospital Ecoville, Curitiba
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Facili - Centro Integrado de Psiquiatria, São Bernardo do Campo
  - BR Trials-Ensaios Clinicos e Consultoria, São Paulo
- Bulgaria (7):
  - ET Dr. Ivo Natsov-AIPSMC in Psychiatry, Cherven Bryag
  - Medical Center Lifemed, Kardzhali
  - DCC Higia, Pazardzhik
  - Medical center Medconsult Pleven OOD, Pleven
  - Mental Health Centre-Prof. N Shipkovenski EOOD, Sofia
  - DCC St. Vrach and St. St. Kuzma and Damian OOD, Sofia
  - UMHAT Alexandrovska EAD, Sofia
- Chile (4):
  - Psicomed Estudios Medicos, Antofagasta
  - Biomedica Research Group, Santiago
  - Especialidades Medicas L y S, Santiago
  - CIC de la Universidad Catolica CICUC, Santiago
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - BRAIN-SOULTHERAPY s.r.o, Kladno
  - AD71 s.r.o, Prague
  - Clinical s.r.o, Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- France (2):
  - Hôpital Lariboisière, Paris
  - Hôpital La Grave, Toulouse
- Italy (2):
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Universitaria OO. RR. S, Salerno
- Mexico (6):
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Neuvo Leon
  - Iecsi S.C., Monterrey, Nuevo León
  - Neurociencias Estudios Clinicos, Culiacán, Sinaloa
  - Centro para el Des de la Med y de Asist Med Esp SC, Culiacán, Sinaloa
  - Hospital Universitario de Saltillo, Coahuila
  - BIND Investigaciones S.C., San Luis Potosí City
- Serbia (6):
  - Clinical Center Dr Dragisa Misovic Dedinje, Belgrade
  - Special Hospital for Psychiatric Diseases, Gornja Toponica
  - Special Hospital for Psychiatric Diseases Kovin, Kovin
  - Jovanovic University Clinical Centre of Kragujevac, Kragujevac
  - Petrovic University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
- South Korea (5):
  - The Catholic University of Korea, Seoul, Republic of Korea
  - Inha University Hospital, Incheon
  - Hanyang University Seoul Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
- Spain (2):
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Provincial de Zamora, Zamora
- Taiwan (3):
  - Kaohsiung Municipal Ta-Tung Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City

IPD SHARING:
Plan to Share IPD: No